CLINICAL TRIAL: NCT00738647
Title: Assessment of a New Resin-based Composite Restorative Material
Brief Title: Assessment of a New Resin-based Composite Filling Material
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Filtek
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-11

CONDITIONS: Caries; Restoration Defects
Keywords: Filling materials; Restorative materials; clinical trial; Resin based composite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ceram X (Active Comparator): Fillings made with a traditional composite material (Ceram X)
  Interventions: Procedure: Tooth restorations with composite
- Filtek Silorane (Experimental): Fillings made with a new composite material (Filtek silorane)
  Interventions: Procedure: Tooth restorations with composite

INTERVENTIONS:
Procedure: Tooth restorations with composite — The cavity is excavated and filled according to the guidelines for composite restorations

SUMMARY:
Evaluation of a new resin-based composite material.

Amalgam and composite are the most commonly used restorative materials in dentistry. Due to the toxicity of mercury and the subsequent environmental problems, the search for alternatives continues and search into new composite restorative materials intensifies. The presently available composites have improved, but shrinkage of the composite during the curing procedure is still a clinical problem. A new composite restorative material has among other advantages demonstrated lower shrinkage in laboratory studies, due to a new formulation of the material.

This project aims to study the clinical performance of this new composite compared to a commonly used composite restoration material. 72 patients (158 teeth) are allocated to the project which is carried out at the School of dentistry, University of Aarhus, Denmark.

DETAILED DESCRIPTION:
This project aims to study the clinical performance of a new composite restoration material (Filtek Silorane®) compared to a conventional composite restoration material (Ceram X®).

Amalgam and composite are the most commonly used restorative materials, with the number of composite restorations increasing over the past 20 years. Composite restorative materials have improved considerably over the years. They have almost reached the same resistance to wear as amalgam, and are as a consequence now also used for molar restorations.

The main reasons for replacing composite restorations are fractures and caries associated with the restorations.

To reduce the risk of caries a new composite material Filtek Silorane® with reduced polymerization shrinkage has been developed.

Extensive laboratory studies have been performed on the new material, but the clinical attributes have yet to be disclosed.

The study will be carried out as a randomized, double blinded, longitudinal study, with assessment of the restorations after one year.

The project includes 72 patients, 158 teeth. Most of the patients have been recruited from the Treatment Planning Clinic at the dental school in Aarhus. After giving their consent to take part in the study, the teeth are randomized into two treatment groups. Multi surface restorations of both upper and lower molars and premolars are performed

The treatment procedure is:

The patients are offered local anesthetic before treatment start. The cavity is excavated and filled according to the guidelines for composite restorations. An impression of the cavity is taken before and after it has been filled. After treatment bw-radiographs are taken.

The control procedure is:

The restoration is evaluated according to marginal adaptation, cavo surface marginal discoloration, approximal contact, fractures, caries associated with restorations and postoperative hypersensitivity. The controls will take place after three weeks and one year.

ELIGIBILITY:
Inclusion Criteria:

* Patients registered for treatment with a posterior multi surface composite restoration.

Exclusion Criteria:

* Poor oral hygiene or teeth needing endodontic treatment.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2007-05; Primary Completion 2018-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Marginal Adaptation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Malene Schmidt, DDS, Principal Investigator — Department of Paediatric Dentistry, School of Dentistry, University of Aarhus